CLINICAL TRIAL: NCT02121132
Title: Establishment of the Pediatric Obesity Weight Evaluation Registry (POWER): A Prospective Pilot Project of Children and Adolescents Presenting for Weight Management
Brief Title: Pediatric Obesity Weight Evaluation Registry (POWER) Study
Acronym: POWER
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Helen DeVos Children's Hospital (Other); Mayo Clinic (Other); Duke University (Other); National Association of Children's Hospitals and Related Institutions (NACHRI) (Unknown); Milton S. Hershey Medical Center (Other); University of New Mexico (Other); University of Illinois College of Medicine at Peoria (Other); Children's Hospital Los Angeles (Other); Connecticut Children's Medical Center (Other); The Children's Hospital of San Antonio (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); Children's Mercy Hospital Kansas City (Other); Arkansas Children's Hospital Research Institute (Other); Florida Hospital for Children (Other); UCSF Benioff Children's Hospital Oakland (Other); University of Oklahoma (Other); MaineHealth (Other); Seattle Children's Hospital (Other); Eastern Maine Medical Center (Other); University of Florida (Other); University of California, Los Angeles (Other); Gramercy Pediatrics (Other); St. Louis Children's Hospital (Other); Dartmouth-Hitchcock Medical Center (Other); University of Alabama at Birmingham (Other); University of Tulsa (Other); Northern Arizona Healthcare (Other); University of Kentucky (Other); Arnold Palmer Hospital for Children (Other); The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-7127
Record Dates: First submitted 2014-04-21; First posted 2014-04-23 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Overweight; Obesity
Keywords: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment

SUMMARY:
The main objective of this study is to establish a national pediatric obesity registry known as POWER (Pediatric Obesity Weight Evaluation Registry). This registry will contain clinical data from individual comprehensive pediatric weight management programs around the United States for overweight and obese youth.

DETAILED DESCRIPTION:
All patients 18 years of age or younger who have completed an initial medical assessment between March 1, 2014 through April 30, 2020 will be approached for this study.

Data from individual follow up visits or group intervention sessions, depending on the program design of each institution, will be collected through October 31, 2020. The data included in this study will be collected during routine medical care. Information that could identify a participant will be removed from the data. Data will be entered into a secure database called Medidata Rave® CDMS. This database will be managed by the Data Coordinating Center (DCC) at Cincinnati Children's Hospital Medical Center (CCHMC).

The DCC will combine all the data from each site. Additional data cleaning and data quality monitoring will be performed. Combined datasets for analysis will be provided by the DCC in a format agreed upon by the POWER Governance Board. Data will be stored in a secure and protected format and will not include any written or electronic protected health information (PHI/EPHI). The DCC will store the data on a secure server.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or younger
* overweight or obese patient
* initial medical evaluation in a pediatric weight management program between March 1, 2014-April 30, 2020.

Exclusion Criteria:

* no exclusion criteria

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will be overweight and obese patients (18 years of age or younger) who are seen for an initial medical evaluation in a pediatric weight management program from March 1, 2014 through April 30, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 4276 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Assess Patient Response to Weight Management Program | 2 years
  This is a composite outcome measure that will be measured with changes in patient weight and BMI, fasting lipid profile, liver enzymes, fasting glucose and insulin, hemoglobin A1C and blood pressure.

SECONDARY OUTCOMES:
Measure Program Retention | 2 years
  This will be measured by the number of visits and days that occur after the initial medical evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Shelley Kirk, PhD, RD, LD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (38):
- United States (38):
  - Fit Kids of Arizona at Northern Arizona Healthcare, Cottonwood, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - University of Florida Health Science Center, Jacksonville, Florida
  - AdventHealth, Orlando, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - St. Luke's Children's Hospital, Boise, Idaho
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Advocate Children's Hospital, Park Ridge, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Riley Children's Hospital - IU Health, Indianapolis, Indiana
  - Our Lady of the Lake, Baton Rouge, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Medical Center - Barbara Bush Children's Hospital, Portland, Maine
  - University of Michigan C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - University of Minnesota Amplatz Children's Hospital, Minneapolis, Minnesota
  - Mayo Clinic in Minnesota, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Children's Hospital and Medical Center Omaha, Omaha, Nebraska
  - University of New Mexico Children's Hospital, Albuquerque, New Mexico
  - Duke Children's Hospital & Health Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - The Medical University of South Carolina, Charleston, South Carolina
  - Dell Children's Medical Center, Austin, Texas
  - Children's Medical Center at UT Southwestern, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - VCU Health, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Marshfield Clinic, Wisconsin Rapids, Wisconsin

REFERENCES:
- [Background] Ogden CL, Carroll MD, Curtin LR, Lamb MM, Flegal KM. Prevalence of high body mass index in US children and adolescents, 2007-2008. JAMA. 2010 Jan 20;303(3):242-9. doi: 10.1001/jama.2009.2012. Epub 2010 Jan 13. PMID 20071470
- [Background] Barlow SE, Dietz WH. Obesity evaluation and treatment: Expert Committee recommendations. The Maternal and Child Health Bureau, Health Resources and Services Administration and the Department of Health and Human Services. Pediatrics. 1998 Sep;102(3):E29. doi: 10.1542/peds.102.3.e29. PMID 9724677
- [Background] Daniels SR, Greer FR; Committee on Nutrition. Lipid screening and cardiovascular health in childhood. Pediatrics. 2008 Jul;122(1):198-208. doi: 10.1542/peds.2008-1349. PMID 18596007
- [Background] Krebs NF, Himes JH, Jacobson D, Nicklas TA, Guilday P, Styne D. Assessment of child and adolescent overweight and obesity. Pediatrics. 2007 Dec;120 Suppl 4:S193-228. doi: 10.1542/peds.2007-2329D. PMID 18055652
- [Background] National High Blood Pressure Education Program Working Group on High Blood Pressure in Children and Adolescents. The fourth report on the diagnosis, evaluation, and treatment of high blood pressure in children and adolescents. Pediatrics. 2004 Aug;114(2 Suppl 4th Report):555-76. No abstract available. PMID 15286277
- [Background] Schwimmer JB, Deutsch R, Rauch JB, Behling C, Newbury R, Lavine JE. Obesity, insulin resistance, and other clinicopathological correlates of pediatric nonalcoholic fatty liver disease. J Pediatr. 2003 Oct;143(4):500-5. doi: 10.1067/S0022-3476(03)00325-1. PMID 14571229
- [Background] Barlow SE; Expert Committee. Expert committee recommendations regarding the prevention, assessment, and treatment of child and adolescent overweight and obesity: summary report. Pediatrics. 2007 Dec;120 Suppl 4:S164-92. doi: 10.1542/peds.2007-2329C. PMID 18055651
- [Background] Spear BA, Barlow SE, Ervin C, Ludwig DS, Saelens BE, Schetzina KE, Taveras EM. Recommendations for treatment of child and adolescent overweight and obesity. Pediatrics. 2007 Dec;120 Suppl 4:S254-88. doi: 10.1542/peds.2007-2329F. PMID 18055654
- [Derived] Christison A, Tucker J, King E, Sweeney B, Cuda S, Frank M, Kirk S. Treating Children and Adolescents With Obesity: Characteristics of Success. Child Obes. 2024 Sep;20(6):416-424. doi: 10.1089/chi.2023.0083. Epub 2023 Nov 15. PMID 37971786
- [Derived] Kumar S, King EC, Christison AL, Kelly AS, Ariza AJ, Borzutzky C, Cuda S, Kirk S; POWER Work Group. Health Outcomes of Youth in Clinical Pediatric Weight Management Programs in POWER. J Pediatr. 2019 May;208:57-65.e4. doi: 10.1016/j.jpeds.2018.12.049. Epub 2019 Mar 8. PMID 30853195
- [Derived] Gross AC, Kaizer AM, Kelly AS, Rudser KD, Ryder JR, Borzutzky CR, Santos M, Tucker JM, Yee JK, Fox CK; POWER Work Group. Long and Short of It: Early Response Predicts Longer-Term Outcomes in Pediatric Weight Management. Obesity (Silver Spring). 2019 Feb;27(2):272-279. doi: 10.1002/oby.22367. PMID 30677263